CLINICAL TRIAL: NCT06833697
Title: A Comparative Study of Erector Spinae Plane Block and Serratus Posterior Superior Intercostal Plane Block on Postoperative Opioid Consumption Following Breast and Axillary Dissection Surgery: A Randomized Controlled Trial
Brief Title: A Comparative Study of Erector Spinae Plane Block and Serratus Posterior Superior Intercostal Plane Block on Postoperative Opioid Consumption Following Breast and Axillary Dissection Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Burak Omur, Assistant Professor, Medipol University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: breast ESP vs SPSİP
Record Dates: First submitted 2025-01-13; First posted 2025-02-19 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Breast Surgery; Erector Spinae Plane Block; Serratus Posterior Superior Intercostal Plane Block
Keywords: Breast surgery; Postoperative pain; Erector spinae plane block; Serratus Posterior Superior Intercostal Plane Block; Opioid consumption; Ultrasound-guided nerve block
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (No Intervention): Patients will not receive any nerve block
- ESPB group (Experimental): Patients will receive an erector spinae plane block.
  Interventions: Procedure: erector spinae plane block; Drug: 0.25% bupivacaine
- SPSIP group (Experimental): Patients will receive a serratus posterior superior intercostal plane block
  Interventions: Procedure: serratus posterior superior intercostal plane block; Drug: 0.25% bupivacaine

INTERVENTIONS:
Procedure: erector spinae plane block — the ESP block will be administered after surgery but before the patient is awakened, under sterile conditions and ultrasound guidance.
  Patient Positioning: The patient will be placed in the lateral position with the surgical side up, and a sterile ultrasound probe cover will be used.
  Ultrasound Imaging: A high-frequency (11-12 MHz) linear probe will be placed transversely at the T5 thoracic vertebra.
  Anatomy Identification: The erector spinae muscle and transverse processes will be visualized.
  Needle Insertion: Using an in-plane technique, the needle will be advanced to the transverse process.
  Injection: After confirming the needle position with 1-2 mL saline, 30 mL of 0.25% bupivacaine will be injected between the erector spinae muscle and transverse process, with spread monitored via ultrasound.
  Arms: ESPB group
Procedure: serratus posterior superior intercostal plane block — In Group 3, SPSIP block will be administered after surgery but before the patient is awakened, under sterile conditions and ultrasound guidance.
  Patient Positioning: The patient will be placed laterally with the surgical side up, using a sterile ultrasound probe cover.
  Ultrasound Imaging: A high-frequency (11-12 MHz) linear probe will be positioned sagittally at the scapula's upper corner to visualize the rhomboid major, trapezius, serratus posterior superior muscles, and the third rib.
  Anatomy Identification: The third rib and serratus posterior superior muscle will be identified.
  Needle Insertion: Using an in-plane technique, the needle will be advanced between the serratus posterior superior muscle and the third rib.
  Injection: After confirming the needle position with 1-2 mL saline, 30 mL of 0.25% bupivacaine will be injected into the space, with spread monitored via ultrasound.
  Arms: SPSIP group
Drug: 0.25% bupivacaine — 0.25% bupivacaine
  Arms: ESPB group; SPSIP group

SUMMARY:
Breast surgery is one of the most common surgical procedures worldwide. Pain after surgery is an important issue because it affects recovery and mobility. It can also increase the risk of breathing problems.

Although opioids are effective for pain relief, they can cause side effects like nausea, vomiting, and breathing difficulties. These side effects can negatively impact patients and their recovery. Reducing opioid use is important for ensuring patient safety and improving the recovery process.

To manage pain after breast surgery, two types of nerve blocks can be used: the erector spinae plane block (ESPB) and the serratus posterior superior intercostal plane block (SPSIP). Both methods are effective for providing pain relief after surgery. However, there are not enough studies comparing which method is better.

Purpose of the Study: The main aim of this study is to evaluate the effect of ultrasound-guided ESPB and SPSIP blocks on opioid use after breast surgery. Additionally, we will compare opioid-related side effects (like nausea, vomiting, and breathing problems) and pain levels measured with the NRS (Numeric Rating Scale) between the two groups.

DETAILED DESCRIPTION:
Introduction Breast surgery is one of the most commonly performed surgical procedures worldwide. Postoperative pain is a significant issue as it impacts recovery and mobilization. Additionally, postoperative pain increases the risk of respiratory complications.

Although opioid analgesics are effective in controlling pain, their side effects, such as nausea, vomiting, and respiratory depression, can lead to undesirable outcomes. Reducing opioid use is critical for both patient safety and improving the quality of recovery.

For managing postoperative pain following breast surgery, the erector spinae plane block (ESPB) and the more recently introduced serratus posterior superior intercostal plane block (SPSIP) have been utilized. Both techniques have been effectively used for analgesia in patients undergoing breast surgery.

However, there is insufficient evidence in the literature comparing the efficacy of these two techniques in this context.

Aim of the Study The primary aim of this study is to evaluate the effect of ultrasound-guided ESPB and SPSIP blocks on postoperative opioid consumption following breast surgery. Additionally, the secondary aim is to compare opioid-related side effects (e.g., nausea, vomiting, respiratory depression) and postoperative NRS (Numerical Rating Scale) pain scores between the groups.

Materials and Methods This prospective, randomized controlled trial will be conducted at Medipol Mega University Hospital on patients undergoing breast surgery and axillary lymph node dissection. The study aims to evaluate the effects of ESPB and SPSIP applications on postoperative opioid consumption and pain management. Written and verbal informed consent will be obtained from all participants prior to the study.

Patient Selection Patients aged 18-80 years, classified as ASA (American Society of Anesthesiologists) physical status I-III, and scheduled for breast surgery with axillary lymph node dissection will be included. Patients with a history of allergies, known allergy to local anesthetics, pregnancy, or psychiatric or neurological disorders will be excluded.

Group Allocation

Patients will be randomized into three groups:

Group 1 (Control group): Patients will not receive any nerve block. Group 2 (ESPB group): Patients will receive an erector spinae plane block. Group 3 (SPSIP group): Patients will receive a serratus posterior superior intercostal plane block.

Anesthesia Management All patients will receive routine anesthesia protocols. After entering the operating room, patients will be monitored with electrocardiography, peripheral oxygen saturation (SpO₂), and non-invasive blood pressure. Premedication with 2 mg intravenous midazolam will be administered.

Anesthesia induction will include 2-2.5 mg/kg IV propofol, 1-1.5 µg/kg IV fentanyl, and 0.6 mg/kg IV rocuronium, followed by intubation. Patients will be ventilated with a 50% oxygen-air mixture. Maintenance of anesthesia will be achieved with intermittent doses of midazolam, fentanyl, and rocuronium. Ventilator settings will include a tidal volume of 6-8 mL/kg and an end-tidal CO₂ of 30-35 mmHg.

All patients will receive 1 g intravenous paracetamol and 100 mg intravenous tramadol 30 minutes before the end of surgery. To prevent postoperative nausea and vomiting, 4 mg intravenous ondansetron will be administered.

Erector Spinae Plane Block Procedure In Group 2, ESPB will be performed following the surgical procedure but before the patient is awakened. The block will be performed under sterile conditions using ultrasound guidance.

Patient Positioning and Preparation: The patient will be positioned laterally with the surgical side up. A sterile ultrasound probe cover will be used.

Ultrasound Imaging: A high-frequency (11-12 MHz) linear ultrasound probe will be placed transversely over the T5 thoracic vertebra.

Identification of Anatomy: The erector spinae muscle and transverse processes will be identified.

Needle Insertion: Using an in-plane technique, the block needle will be advanced to the transverse process.

Injection Confirmation: After confirming the needle position with a 1-2 mL saline injection, 30 mL of 0.25% bupivacaine will be injected between the erector spinae muscle and the transverse process. Spread of the local anesthetic will be monitored via ultrasound.

Serratus Posterior Superior Intercostal Plane Block Procedure In Group 3, SPSIPB will also be performed following the surgical procedure but before the patient is awakened. The block will be performed under sterile conditions using ultrasound guidance.

Patient Positioning and Preparation: The patient will be positioned laterally with the surgical side up. A sterile ultrasound probe cover will be used.

Ultrasound Imaging: A high-frequency (11-12 MHz) linear ultrasound probe will be placed sagittally at the upper corner of the scapula. The rhomboid major, trapezius, serratus posterior superior muscles, and the third rib will be visualized.

Identification of Anatomy: The third rib and serratus posterior superior muscle will be identified.

Needle Insertion: Using an in-plane technique, the block needle will be advanced between the serratus posterior superior muscle and the third rib.

Injection Confirmation: After confirming the needle position with a 1-2 mL saline injection, 30 mL of 0.25% bupivacaine will be injected into the space between the serratus posterior superior muscle and the third rib. Spread of the local anesthetic will be monitored via ultrasound.

Postoperative Assessment Pain levels will be assessed during the first 24 hours postoperatively. Patients will routinely receive 1,000 mg paracetamol three times daily. Pain scores will be evaluated using the Numerical Rating Scale (NRS), where 0 indicates "no pain" and 10 indicates "worst pain imaginable."

Pain scores at rest and during mobilization will be recorded at the recovery unit, as well as at 3, 6, 12, 18, and 24 hours postoperatively. If the NRS score is ≥4, 1 mg/kg IV tramadol will be administered as rescue analgesia. The total amount of rescue analgesic used, postoperative opioid consumption, and side effects such as nausea, vomiting, itching, and complications like hematoma will be documented.

ELIGIBILITY:
Inclusion Criteria:

* aged 18-80 years
* Classified as ASA (American Society of Anesthesiologists) physical status I-III
* Scheduled for breast surgery with axillary lymph node dissection

Exclusion Criteria:

* Patients with a history of allergies
* allergic to local anesthetics
* pregnant women
* psychiatric or neurological disorders

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2025-01-27 (Actual); Primary Completion 2025-08-01 (Actual); Study Completion 2025-09-01 (Actual)

PRIMARY OUTCOMES:
tramadol consumption | irst 24 hours after the operation
  Total tramadol consumption (mg) in the first 24 hours after surgery.

SECONDARY OUTCOMES:
NRS (Numerical Rating Scale) pain scores | first 24 hours after the operation
  NRS (0-10) scores will be measured at 3, 6, 12, 18, and 24 hours during both rest and mobilization in the postoperative period.
opioid-related side effects (such as nausea, vomiting, respiratory depression) | first 24 hours after the operation
  The incidence of opioid-related side effects (e.g., nausea, vomiting, respiratory depression) will be recorded and compared between groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Medipol University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
only IPD used in the results publication

REFERENCES:
- [Background] Cortes-Flores AO, Jimenez-Tornero J, Morgan-Villela G, Delgado-Gomez M, Zuloaga-Fernandez Del Valle CJ, Garcia-Renteria J, Rendon-Felix J, Fuentes-Orozco C, Macias-Amezcua MD, Ambriz-Gonzalez G, Alvarez-Villasenor AS, Urias-Valdez D, Chavez-Tostado M, Contreras-Hernandez GI, Gonzalez-Ojeda A. Effects of preoperative dexamethasone on postoperative pain, nausea, vomiting and respiratory function in women undergoing conservative breast surgery for cancer: Results of a controlled clinical trial. Eur J Cancer Care (Engl). 2018 Jan;27(1). doi: 10.1111/ecc.12686. Epub 2017 May 4. PMID 28474341
- [Background] Ciftci B, Ekinci M, Yildiz Y. Erector Spinae Plane Block for a Patient who Underwent Both Bilateral Mastectomy and Right Video-Assisted Thoracic Surgery. Turk J Anaesthesiol Reanim. 2020 Apr;48(2):170-171. doi: 10.5152/TJAR.2019.01205. Epub 2019 Nov 11. No abstract available. PMID 32259153
- [Background] Ciftci B, Alver S, Ahiskalioglu A, Bilal B, Tulgar S. Serratus posterior superior intercostal plane block for breast surgery: a report of three cases, novel block and new indication. Minerva Anestesiol. 2023 Nov;89(11):1054-1056. doi: 10.23736/S0375-9393.23.17432-3. Epub 2023 Jun 1. No abstract available. PMID 37272274